CLINICAL TRIAL: NCT06587126
Title: Assessing the Feasibility of Home Nighttime Cough Monitoring in Children with Cystic
Brief Title: Feasibility of Cough Monitoring in Children
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0382
Record Dates: First submitted 2024-08-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Children with Cystic Fibrosis: Childrens ages 1-18 with a diagnosis of CF based on 2 known cystic fibrosis transmembrane conductance regulator (CFTR) mutations and/or sweat chloride >60 mmol/L, thought to be clinically stable at the time of study consent.
  Interventions: Device: Curie Artificial Intelligence (AI) cough monitor
- Healthy Controls: Children ages 1-18 with no underlying respiratory of cardiac conditions including chronic cough, CF, asthma, obstructive sleep apnea, or congenital heart disease thought to cause chronic nighttime symptoms.
  Interventions: Device: Curie Artificial Intelligence (AI) cough monitor

INTERVENTIONS:
Device: Curie Artificial Intelligence (AI) cough monitor — All patients are given nighttime cough monitors for home use for 3-4 months

SUMMARY:
Cystic fibrosis (CF) is a disease characterized by chronic airway infection and impaired mucociliary clearance, which predisposes those affected to recurrent pulmonary exacerbations (PEx) and progressive decline in lung function. Treatment with elexacaftor/tezacaftor/ivacaftor (ETI) results in decreases in patient-reported cough and PEx. Despite this, increased cough remains the most common symptom associated with acute PEx and worsening lung disease. Cough frequency was historically difficult to measure due to reliance on human input. Recent advances in audio capture and signal processing have made automated cough detection possible. As a result there's been a surge in development of portable cough monitors, as cough is increasingly recognized as a measurable parameter of respiratory disease. The majority of cough monitors have been designed for use in adults, and little is known about the practicality of collecting cough data in the pediatric population. In this study investigators aim to assess the feasibility of using an in-home device to capture nighttime cough frequency in children with and without CF. Investigators plan to compare nighttime cough frequency between children with and without CF and, among children with CF, and determine the association between cough frequency and baseline lung function. Additionally, investigators aim to evaluate the changes in nighttime cough frequency in relationship to respiratory symptom scores surrounding clinician diagnosed pulmonary exacerbations. This study will provide important preliminary data needed for a larger study assessing the utility of home cough monitoring for clinical care and for use of cough as a clinical outcome measure in research studies.

ELIGIBILITY:
Inclusion Criteria for Children with Cystic Fibrosis

* Diagnosis of CF based on 2 known CFTR mutations and/or sweat chloride > 60 mmol/L
* Ages 1-18 years of age
* Clinically stable at the time of consent

Exclusion Criteria

* Use of nocturnal positive pressure or supplemental oxygen
* Shared bedroom with sibling
* Use of oral or IV antibiotics within the past 2 weeks except for chronic azithromycin use
* Shared custody (i.e., the participant is splitting time between time households)

Inclusion Criteria for Healthy Controls

* Ages 1-18

Exclusion Criteria:

* Shared bedroom with sibling
* Underlying chronic respiratory or cardiac conditions including chronic cough, CF, asthma, obstructive sleep apnea, or congenital heart disease or other condition felt by the investigator to cause chronic nighttime symptoms
* Shared custody (i.e., the participant is splitting time between time households)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: See inclusion and exclusion criteria for both groups above. Our aim to recruit 20 participants in each cohort.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using an in-home cough monitoring device | Through study completion, an average of 3 months
  Percent of nights over the study period during which 4 or more hours of analyzable data are collected over study period

SECONDARY OUTCOMES:
Comparison of nighttime cough between participants with CF and healthy controls | Through study completion, an average of 3 months
  Average cough seconds per hour per night over the study period
Comparison of nighttime cough in children with CF during clinician diagnosed pulmonary exacerbations | 7 days
  Assess for changes in cough frequency before and after diagnosis of pulmonary exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Lilah Melzer, DO, Principal Investigator — Children's Hospital Colorado, University of Colorado
Locations (1):
- Children's Hospital of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided